#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for 205184: A single-centre, randomized, double-blind (sponsor-unblinded), placebocontrolled study to evaluate the safety, tolerability and pharmacokinetics of GSK2982772 in repeat oral doses in healthy subjects

Compound Number : GSK2982772

Effective Date : 30-NOV-2018

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205184.
- This RAP is intended to describe the safety, tolerability and PK analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC deliverable).

#### **RAP Author(s):**

| Approver | | Date | Approval<br>Method |
|---|---|---|---|
| Statistics Leade | er (II Clinical Statistics) | 19-NOV-2018 | Email |
| Principal Statis | tician I (Quanticate) | 15-NOV-2018 | Email |
| Principal Statis | tician (II Clinical Statistics) | 13-NOV-2018 | Email |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Clinical Development Scientist, GCSD II | 16-NOV-2018 | Email |
| PPD Clinical Investigational Lead, iiTA | 15-NOV-2018 | Email |
| PPD Director, CPMS | 16-NOV-2018 | Email |
| Project Physician Lead, iiTA | 21-NOV-2018 | Email |
| Senior Medical Director, GCSP SERM | 19-NOV-2018 | Email |
| Data Quality Lead, Global Clinical & Data Operations | 19-NOV-2018 | Email |
| Principal Programmer, II Clinical Programming | 15-NOV-2018 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Senior Statistics Director, II Clinical Statistics | 28-NOV-2018 | CARS<br>e-Signature |
| Programming Manager, II Clinical Programming | 30-NOV-2018 | CARS<br>e-Signature |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 5 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION | 5<br>5 |
| 3. | PLANI<br>3.1.<br>3.2. | NED ANALYSES Interim Analyses Final Analyses | 9 |
| 4. | ANAL`<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS Study Treatment & Sub-group Display Descriptors Baseline Definitions Multicentre Studies Examination of Covariates, Other Strata and Subgroups Multiple Comparisons and Multiplicity Other Considerations for Data Analyses and Data Handling Conventions | 11<br>12<br>12 |
| 6. | SAFE <sup>1</sup><br>6.1.<br>6.2.<br>6.3. | TY ANALYSES Adverse Events Analyses Clinical Laboratory Analyses Other Safety Analyses | 14<br>14 |
| 7. | STUD<br>7.1. | OY POPULATION ANALYSESOverview of Planned Study Population Analyses | |
| 8. | PHAR<br>8.1. | RMACOKINETIC ANALYSES Primary Pharmacokinetic Analyses 8.1.1. Endpoint / Variables 8.1.1.2. Derived Pharmacokinetic Parameters 8.1.2. Summary Measure 8.1.3. Population of Interest 8.1.4. Strategy for Intercurrent (Post-Randomization) Events Secondary Pharmacokinetic Analyses 8.2.1. Endpoint / Variables 8.2.1.1. Drug Concentration Measures | 16<br>16<br>16<br>17<br>17<br>17 |
| 9. | REFE | RENCES | 18 |
| 10 | APPF | NDICES | 19 |

#### CONFIDENTIAL

| 2 | ი51 | ۱۵/ |
|---|-----|-----|

| 10.1. | Appendix | x 1: Protocol Deviation Management | 19 |
|--------|----------|----------------------------------------------------|----|
| 10.2. | Appendix | x 2: Schedule of Activities | 20 |
| | 10.2.1. | Protocol Defined Schedule of Events | 20 |
| | | 10.2.1.1. Part A (Cohort 1) | |
| | | 10.2.1.2. Part B (Cohorts 2-5) | 23 |
| 10.3. | Appendix | x 3: Assessment Windows | |
| | 10.3.1. | Definitions of Assessment Windows for Analyses | |
| 10.4. | Appendix | x 4: Study Phases and Treatment Emergent Adverse | |
| | | | 42 |
| | 10.4.1. | Study Phases | |
| | | 10.4.1.1. Study Phases for Concomitant Medications | |
| | 10.4.2. | Treatment Emergent Flag for Adverse Events | |
| 10.5. | | x 5: Data Display Standards & Handling Conventions | |
| | 10.5.1. | Reporting Process | |
| | 10.5.2. | Reporting Standards | |
| | 10.5.3. | Reporting Standards for Pharmacokinetic | |
| 10.6. | | x 6: Derived and Transformed Data | |
| | 10.6.1. | General | |
| | 10.6.2. | Study Population | |
| | 10.6.3. | Safety | |
| 10.7. | | x 7: Reporting Standards for Missing Data | |
| | 10.7.1. | Premature Withdrawals | 47 |
| | 10.7.2. | Handling of Missing Data | |
| | | 10.7.2.1. Handling of Missing and Partial Dates | |
| 10.8. | Appendix | x 8: Values of Potential Clinical Importance | |
| | 10.8.1. | Laboratory Values | |
| | 10.8.2. | • | |
| | 10.8.3. | Vital Signs | |
| 10.9. | | x 9: Abbreviations & Trade Marks | |
| | 10.9.1. | | |
| | 10.9.2. | | |
| 10.10. | Appendix | x 10: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | 54 |
| | | Safety Tables | |
| | | Safety Figures | |
| | 10.10.7. | Pharmacokinetic Tables | 65 |
| | | Pharmacokinetic Figures | |
| | 10.10.9. | ICH Listings | 68 |
| | | Non-ICH Listings | |
| 10.11. | | x 11: Example Mock Shells for Data Displays | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 205184:

| Revision Chronology: | | |
|----------------------|-------------|--------------------------|
| 2017N326600_00 | 31-JUL-2017 | Original |
| 2017N326600_01 | 07-DEC-2017 | Amendment 01 |
| 2017N326600_02 | 15-FEB-2018 | Amendment 02 |
| 2017N326600_03 | 26-FEB-2018 | Republished Amendment 02 |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| An interim analysis may be performed during the study on completed cohorts in Part A and Part B of the study to aid internal decision making only. The RAP will describe the planned interim analyses in greater detail. | No formal IA will be conducted during the study. | The DEC make decisions on proceeding to higher dose strengths based on assessment of safety, tolerability and pharmacokinetic data at the preceding dose only. |
| Protocol Section 10.3 references an 'Enrolled population'. | RAP uses the 'Randomised Population'. | The population was renamed to match the current IDSL guidance. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To investigate the safety and tolerability of repeat doses of GSK2982772 in healthy subjects. | <ul> <li>Adverse events.</li> <li>Clinical laboratory values (clinical chemistry, haematology and urinalysis).</li> <li>Vital sign measurements (blood pressure, heart rate, respiratory rate and body temperature).</li> <li>Physical examinations.</li> <li>12-Lead ECG monitoring.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Secondary Objectives | Secondary Endpoints |
| To characterise the pharmacokinetic (PK) profile of repeat doses of GSK2982772 in healthy subjects. | • A 24 hr profile to be collected on Day 1 of Part A and Day 14 of Part B. On Day 1 of Part B, the PK profile will be evaluated following the first dose only. Derived PK parameters for GSK2982772, including area under the plasma drug concentration versus time curve over 24 hr (AUC <sub>(0-24)</sub> ) and AUC over each dose interval (i.e. AUC <sub>(0-7)</sub> , AUC <sub>(7-14)</sub> and AUC <sub>(14-24)</sub> for TID and AUC <sub>(0-12)</sub> and AUC <sub>(12-24)</sub> for BID). Maximum observed plasma drug concentration (C <sub>max</sub> ) following each dose, time to maximum observed plasma drug concentration (T <sub>max</sub> ) following each dose, observed trough plasma drug concentrations (C <sub>0</sub> , C <sub>7</sub> , C <sub>14</sub> and C <sub>24</sub> for TID dosing and C <sub>0</sub> , C <sub>12</sub> and C <sub>24</sub> for BID dosing). |
| <ul> <li>To assess the impact of food on the<br/>PK of repeat doses of GSK2982772 in<br/>healthy subjects at steady state</li> </ul> | <ul> <li>Derived PK parameters for GSK2982772, including<br/>AUC<sub>(0-7)</sub>, AUC<sub>(7-14)</sub>, C<sub>max</sub>, after 1<sup>st</sup> dose of day and T<sub>max</sub><br/>after 1<sup>st</sup> dose of day.</li> </ul> |
| To assess potential effect of repeat<br>doses of GSK2982772 on CYP3A4<br>enzyme activity | Plasma 4β-hydroxycholesterol to cholesterol ratio pre-<br>treatment and following 14 days of repeat dosing of<br>GSK2982772. |
| Exploratory Objectives | Exploratory Endpoints |
| To investigate the levels of circulating glucuronide metabolite (M8; GSK3562183) and desmethyl metabolite (M9; GSK2997852) in healthy subjects after single-day and repeat dosing of GSK2982772. | Quantify M8 (GSK3562183) and M9 (GSK2997852) in select plasma PK samples at pre-dose and 2 hr following Day 14 of repeat dosing of GSK2982772. |

#### 2.3. Study Design

#### Overview of Study Design and Key Features Part A - Single-Day Ascending Doses Part B - Repeat Doses Part B - Repeat Doses 1 Day 14 Days 14 Days 3:1 Randomized 3:1 Randomized 9:5 Randomized GSK2982772:Placebo GSK2982772:Placebo GSK2982772:Placebo Cohort 1 Cohort 2 Cohort 3 N=14 N=12 N=12 120 ma TID 120 mg TID (1 Day) followed by, 120 mg TID 14 Days \* 240 mg TID (1 Day) followed by, 14 Days \* 360 mg BID (1 Day) Cohort 4 N=14 240 mg TID 14 Days \* Cohort 5 N=14 360 mg BID 14 Days \*With Food Effect Treatment Design This is a single-centre, randomized, double-blind (sponsor-unblinded), placebo-Features controlled study to evaluate the safety, tolerability and pharmacokinetics of GSK2982772 in repeat oral doses in healthy participants. This study consists of 2 parts: Part A (Cohort 1) – single ascending dose, randomized, placebo-controlled, 3way crossover. Part B (Cohorts 2, 3, 4 and 5) – repeat dose, randomized, placebo-controlled, sequential-group. Time & Refer to Appendix 2: Schedule of Activities **Events** Treatment The study is planned to enrol approximately 66 participants with approximately 12 Assignment participants (9 active, 3 placebo) in Cohorts 1 and 2 (up to approximately 24 in total) and 14 participants (9 active, 5 placebo) in Cohorts 3, 4 and 5 (up to approximately 42 in total). If participants prematurely discontinue the study, additional replacement participants may be randomized in order to guarantee that sufficient participants are treated with GSK2982772 at any given dose before escalating to the following dose. Replacement participants will be assigned to the same treatment sequence (Cohort 1) or treatment (Cohorts 2-5). All participants will be centrally randomized using an Interactive Voice/Web Response System (IVRS/IWRS). Study treatment is dispensed at the study visits summarized in the Schedule of Activities (SoA). Each participant is dispensed blinded study treatment, labelled with his/her unique randomization number, throughout the study. Returned study treatment should not be re-dispensed to the participants.

| Overview of S | tudy Design and Key Features |
|---|---|
| | <ul> <li>In Cohorts 1 and 2, participants will be randomized in a 3:1 ratio to either<br/>GSK2982772 or placebo. In Cohorts 3, 4 and 5, participants will be randomized in a<br/>9:5 ratio to either GSK2982772 or placebo.</li> </ul> |
| | <ul> <li>The randomization will reflect the fact that at least 2 of the 12 participants in Cohorts 1 and 2 and at least 2 of the 14 participants in Cohort 4 and 5 (one participant will receive GSK2982772 and one participant will receive matched-placebo) will be dosed first (on Day 1) in each part to enable dose staggering.</li> <li>In Cohort 1, the participants will be randomized to one of four sequences (ABC, ABP, APC, PBC), where the treatments are: A 120 mg TID B 240 mg TID C 360 mg BID P Placebo</li> <li>Once a treatment allocation number has been assigned to a participant, it cannot be</li> </ul> |
| | reassigned to any other participant. |
| Dosing | <ul> <li>For TID dosing, GSK2982772 or placebo will be administered using a 7hr and 7hr dosing interval in Part A and a 7hr, 7hr and 10hr dosing interval in Part B.</li> <li>For BID dosing, GSK2982772 or placebo will be administered using a 12hr dosing interval.</li> </ul> |
| Interim<br>Analysis | <ul> <li>No interim analyses will be performed.</li> <li>The decision to proceed to higher dose strengths will be made by the Dose Escalation Committee (DEC) based on assessment of safety, tolerability and pharmacokinetic data at the preceding dose.</li> </ul> |

# 2.4. Statistical Hypotheses / Statistical Analyses

- The objectives of this study are to assess the safety and tolerability of single and repeat ascending doses of GSK2982772. No formal hypotheses will be tested.
- An estimation approach will be used to describe pharmacokinetics of GSK2982772, where point estimates and corresponding 90% confidence intervals will be constructed, unless otherwise stated.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No interim analyses will be performed. The decision to proceed to higher dose strengths will be made by the Dose Escalation Committee (DEC) based on assessment of safety, tolerability and pharmacokinetic data at the preceding dose.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects | Comprises of all participant who were screened and allocated a subject number. | <ul><li>Screen Failure</li><li>Population<br/>Analysed.</li></ul> |
| Randomised | <ul> <li>All participants who were randomly assigned to treatment in the study.</li> <li>This population will be based on the treatment the participant was randomized to.</li> </ul> | Age ranges |
| Safety | <ul> <li>Comprises of all randomised participants who received at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject was randomised to.</li> </ul> | <ul><li>All other Study<br/>Population</li><li>Safety</li></ul> |
| Pharmacokinetic | Participants in the 'Safety' population for whom a pharmacokinetic sample was obtained and analysed. | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

Note: All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (Version 4.0, 01 Feb 18)

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group l | Descriptions | |
|---|---|---|---|
| | RandAll NG | Data Displays for Re | eporting |
| Code | Description | Description | Order in<br>TLF |
| Р | Placebo TID Single Dose | Placebo | 1 |
| Q | Placebo BID Single Dose | Placebo | 1 |
| Α | GSK2982772 120 mg TID Single Dose | GSK 120 mg TID | 2 |
| В | GSK2982772 240 mg TID Single Dose | GSK 240 mg TID | 3 |
| С | GSK2982772 360 mg BID Single Dose | GSK 360 mg BID | 4 |
| R | Placebo TID Repeat Dose | Placebo | 1 |
| S | Placebo BID Repeat Dose | Placebo | 1 |
| D | GSK2982772 120 mg TID Repeat Dose | GSK 120 mg TID | 2 |
| Е | GSK2982772 240 mg TID Repeat Dose | GSK 240 mg TID | 3 |
| F | GSK2982772 360 mg BID Repeat Dose | GSK 360 mg BID | 4 |
| G | GSK2982772 Cohort 3 Repeat Dose | GSK 120 mg TID | 2 |
| Н | GSK2982772 Cohort 4 Repeat Dose | GSK 240 mg TID | 3 |
| J | GSK2982772 Cohort 5 Repeat Dose | GSK XX mg TID/BID [1] | 3 or 4 |
| Т | Placebo Cohort 3 Repeat Dose | Placebo | 1 |
| U | Placebo Cohort 4 Repeat Dose | Placebo | 1 |
| V | Placebo Cohort 5 Repeat Dose | Placebo | 1 |

#### NOTES:

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

For Part A, baseline definitions defined in the table are applicable to each treatment period.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing. The mean of triplicate measurements at any given time point will be used as the value for that time point unless otherwise stated.

<sup>[1]</sup> Dose level not required as the study met the PK stopping criteria at the end of Cohort 4.

| Parameter | Study Asses | sments Consid | Baseline Used in | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | | | | |
| Clinical Chemistry/<br>Haematology/<br>Urinalysis | X | Χ | X | Day 1 |
| 12-lead ECG [1] | X | Χ | X | Day 1 |
| Vital Signs | Х | Х | Х | Day 1 |
| C-SSRS (Part B only) | Х | | X | Day -1/Day 1 |
| Pharmacokinetic | | | | |
| PK Concentrations/<br>Parameters | | | Х | Day 1 |

#### NOTES:

### 5.3. Multicentre Studies

This is a single centre study.

# 5.4. Examination of Covariates, Other Strata and Subgroups

There are no covariates, strata or subgroups to be investigated in this study.

# 5.5. Multiple Comparisons and Multiplicity

No adjustments for multiplicity will be required.

<sup>[1]</sup> ECG recordings will be performed in triplicate at screening. Use the mean of the triplicate measurements.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Schedule of Activities |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |
| 10.9 | Appendix 9: Abbreviations & Trademarks |
| 10.10 | Appendix 10: List of Data Displays |
| 10.11 | Appendix 11: Example Mock Shells for Data Displays |

#### 6. SAFETY ANALYSES

All safety analyses will be based on the" Safety" population, unless otherwise specified.

#### 6.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

# 6.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

Additionally, plasma  $4\beta$ -hydroxycholesterol to cholesterol ratio pre-treatment and following 14 days of repeat dosing of GSK2982772 will be summarised and listed.

In addition to GSK Core Data Standards, lipids (Total Cholesterol, Triglycerides, HDL cholesterol, LDL cholesterol and Total Cholesterol/HDL ratio) outside the normal range and percent change in lipids will be summarised. The fasting lipid status will be included in listings.

# 6.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. Suicide risk monitoring including analyses of Colombia Suicide Severity Rating Scale (C-SSRS) will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

## 7. STUDY POPULATION ANALYSES

## 7.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, concomitant medication, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

#### 8. PHARMACOKINETIC ANALYSES

## 8.1. Primary Pharmacokinetic Analyses

### 8.1.1. Endpoint / Variables

#### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Standards for Pharmacokinetic).

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC <sub>(0-24)</sub> | Area under the curve from time zero hours to 24 hours |
| AUC <sub>(0-7)</sub> | Area under the curve from time zero hours to 7 hours (TID only) |
| AUC <sub>(7-14)</sub> | Area under the curve from time 7 hours to 14 hours (TID only) |
| AUC <sub>(14-24)</sub> | Area under the curve from time 14 hours to 24 hours (TID only) |
| AUC <sub>(0-12)</sub> | Area under the curve from time zero hours to 12 hours (BID only) |
| AUC <sub>(12-24)</sub> | Area under the curve from time 12 hours to 24 hours (BID only) |
| Cmax | Maximum observed concentration after 1st, 2nd and 3rd dose in Part A and on Day 14 in Part B |
| Tmax | Time to maximum observed concentration after 1st, 2nd and 3rd dose in Part A and on Day 14 in Part B |
| C <sub>0</sub> | Concentration at zero hours (pre-dose) |
| C <sub>7</sub> | Concentration at 7 hours post-dose (TID only) |
| C <sub>12</sub> | Concentration at 12 hours post-dose (BID only) |
| C <sub>14</sub> | Concentration at 14 hours post-dose (TID only) |
| C <sub>24</sub> | Concentration at 24 hours post-dose |

#### NOTES:

• Additional parameters may be included as required.

#### 8.1.2. Summary Measure

- The PK of TID and BID dosing on Day 1 in Part A will be evaluated. In Part B the comparisons of interest will be:
  - The PK profile following the 1<sup>st</sup> dose of the day following administration in the fed state (standard meal on Day 9 and high fat meal on Day 11) or in the fasted state (Day 14).
  - The pharmacokinetic profile following the 1<sup>st</sup> dose on Day 14 (fasted) and the 1<sup>st</sup> dose on Day 1 (fasted);

Descriptive statistics (n, arithmetic mean, standard deviation [SD] standard error [SE], 95% CI, minimum, median and maximum) will be calculated by treatment for all PK concentrations over time and for the derived PK parameters. In addition, for loge-transformed PK parameter variables geometric mean, 95% CI and %CV<sub>b</sub> (100 \* √ (exp(SD²) -1)) will be provided, where the SD is the standard deviation of log-transformed data

## 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

#### 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

- Study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.
- Withdrawn participants may be replaced in the study. Replacement participants, enrolled will be dosed with the next planned treatment of the withdrawn participant, and they will not receive any treatment that the withdrawn participant has already received with the exception of the need to increase participants numbers to obtain the minimum number of evaluable participants required for interim decisions, and to obtain data in any other treatment that is required for a valid comparison. Replacement participants will receive the required treatments in the same order as planned for the original participant.
- All available data from participants who were withdrawn from the study will be listed
  and all available planned data will be included in summary tables and figures, unless
  otherwise specified.

# 8.2. Secondary Pharmacokinetic Analyses

#### 8.2.1. Endpoint / Variables

#### 8.2.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Standards for Pharmacokinetic).

Descriptive statistics (n, arithmetic mean, standard deviation, standard error, 95% CI, minimum, median and maximum) of circulating glucuronide metabolite (M8; GSK3562183) and des-methyl metabolite (M9; GSK2997852) will be investigated in healthy participants after single-day and repeat dosing of GSK2982772

# 9. REFERENCES

• PKOne and relevant information on Standards for the Transfer and Reporting of PK Data using HARP available within IDSL standards.

## 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.

# 10.2. Appendix 2: Schedule of Activities

## 10.2.1. Protocol Defined Schedule of Events

# 10.2.1.1. Part A (Cohort 1)

| | Screening | St | udy F | Perio | d (Day | s) | Follow-Up | |
|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28 days before Day | -1 | 1 | 2 | 3 | 4 | (No more<br>than 14<br>days post<br>last dose) | Notes |
| Outpatient Visit | Х | | | | | | Х | |
| Admission to Clinical Unit | | Χ | | | | | | |
| Inpatient Stay at Clinical Unit | | | <b>←</b> : | ==X== | <b>-</b> → | | | |
| Discharge from Clinical Unit | | | | | | Χ | | Following completion of all assessments. |
| Informed Consent | X | | | | | | | |
| Inclusion and Exclusion Criteria | X | | | | | | | |
| Demography | X | | | | | | | |
| Full Physical Examination | Х | | | | | | | Additional exams/screens may be performed, or brief exams made full exams, by the Investigator, as deemed necessary (e.g. where safety or laboratory findings indicate). Tests will be conducted within site specified standards. |
| Brief Physical Examination | | Χ | | Х | | Χ | | resis will be conducted within site specified standards. |
| Height | Х | | | | | | | |
| Weight | Х | | | | | | | |
| Drug/Alcohol/Smoking Screen | Х | Χ | | | | | | Tests include alcohol breath test, smoking breath test and urine drug screen. |
| Medical/Medication/Drug/Alcohol History | Х | | | | | | | |
| HIV, Hepatitis B and C Screening | Х | | | | | | | |
| Tuberculosis Test | Х | | | | | | | Conducted at the standard practice of the site. |
| Serum Pregnancy Test (WOCBP only) | X | | | | | | Х | |
| Urine Pregnancy Test (WOCBP only) | | Х | | | | Χ | | |
| Highly effective contraceptive method (WOCBP only) | Х | Х | Х | Х | Х | Х | Х | Must use method for a minimum of 28 days prior to first dose of study medication until the follow-up visit |

| Procedure day before Contraception with male condoms (WOCBP using hormonal contraceptive method and male | to 28 ays<br>ays<br>e Day<br>1) | -1<br>X | 1 | 2 | 3 | 4 | (No more<br>than 14<br>days post | Notes |
|---|---|---|---|---|---|---|---|---|
| (WOCBP using hormonal contraceptive method and male | | Y | | | | | last dose) | |
| subjects with female partners of childbearing potential only) | | ^ | X | Х | Х | X | X | |
| Meals | | X | Χa | х | X | X | | a On Day 1, subjects will fast 8hr overnight prior to dose 1. A breakfast will be served approximately 2hr after dose 1. TID dosing: On Day 1, lunch and dinner will be served between 2 to 3hr prior to doses 2 and 3, respectively. BID dosing: On Day 1, lunch will be served approximately 4 to 5hr after dose 1. Dinner will be served between 2 to 3hr prior to dose 2. A snack may be consumed approximately 2 to 3hr after dose 2. Water is permitted with dosing and at all times. Subjects will receive standardized meals scheduled at the same time in each period. |
| Haem/Chem/Urinalysis Test (Include Liver Chemistries) | х | Χ | Χ | Х | | Χ | Х | Non-fasted samples can be collected on Day -1 and Follow-Up Visit. |
| PK Blood Sampling | | | X | х | | | | TID Dosing: PK samples to be taken pre-dose on Day 1 and then at the following time points post first-dose: 20min, 40min, 1hr, 1hr 30min, 2hr, 3hr, 5hr, 7hr, 7hr 20min, 7hr 40 min, 8hr, 8hr 30min, 9hr, 10hr, 12hr, 14hr, 14hr 20min, 14hr 40 min, 15hr, 15hr 30min, 16hr, 17hr, 19hr, 22hr, 24hr. BID Dosing: PK samples to be taken pre-dose on Day 1 and then at the following time points post first-dose: 20min, 40min, 1hr, 1hr 30min, 2hr, 3hr, 4hr, 6hr, 8hr, 10hr, 12hr, 12hr 20min, 12hr 40min, 13hr, 13hr 30min, 14hr, 15hr, 16hr, 19hr, 22hr, 24hr. Remaining PK plasma samples from Part A may be analysed for metabolite sampling. |
| Neuro. Examination Telemetry | | ←> | ⟨→ | X | ←> | <→ | | TID Dosing: Neurological examinations to be conducted either on Day -1 or pre-dose Day 1 and then at the subsequent time points post first-dose on Day 1: 2hr, 9hr, 16hr, 24hr and 48hr. Then 24 and 48hr after the last dose administered on Day 1. BID Dosing: Neurological examinations to be conducted either on Day -1 or pre-dose Day 1 and then at the subsequent time points post first-dose: 2hr, 14hr, 24hr and 48hr. Then 24 and 48 hr after the last dose administered on Day 1. Continuous at least 24hr post-evening dose. Initiate at least 15 min. prior to dosing. |

| | Screening | S | tudy F | Perio | d (Day | /s) | Follow-Up | |
|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days<br>before Day<br>1) | -1 | 1 | 2 | 3 | 4 | (No more<br>than 14<br>days post<br>last dose) | Notes |
| 12-Lead ECG | X | Х | Т | Х | <b>←</b> > | <b>&lt;</b> > | | Vital signs to include HR, BP, temperature and respiration rate. <u>TID Dosing:</u> 12-Lead ECG and Vital Signs to be conducted on Day -1 and pre-dose on |
| Vital Signs | Х | Х | Т | Х | €) | ⟨→ | Х | Day 1 and then at the subsequent time points post first-dose: 40min, 2hr, 4hr, 7hr (pre-2 <sup>nd</sup> dose), 9hr, 14hr (pre-3 <sup>rd</sup> dose), 16hr, 24hr and 48hr. Then 24 and 48hr after the last dose administered on Day 1. BID Dosing: 12-Lead ECG and Vital Signs to be conducted on Day -1 and pre-dose on Day 1 and then at the subsequent time points post first-dose: 40 min, 2hr, 4hr, pre-2 <sup>nd</sup> dose, 12hr 20 min, 14hr, 24hr and 48 hr. Then 24 and 48hr after the last dose administered on Day 1. T = Triplicate. |
| Randomization | | , | Χ | | | | | Randomization can occur on either Day -1 or Day 1. |
| Study Treatment | | | Xp | | | | | <ul> <li><u>TID dosing:</u> GSK2982772 or placebo will be administered using a 7hr, 7hr dosing interval.</li> <li><u>BID dosing:</u> GSK2982772 or placebo will be administered using a 12hr dosing interval.</li> </ul> |
| Pharmacogenetic Sample (PGx) | | | х | | | | | A PGx blood sample is collected at the Day 1 visit, after the subject has been randomized and provided informed consent for genetic research. If the sample is not collected at the Day 1 visit, it can be collected at any time during the study after randomization. |
| AE Review | | <b>←</b> : | | ==X= | ==== | => | Χ | |
| SAE Review | | <b>←</b> : | | ==X= | ==== | => | X | |
| Concomitant Medication Review | X | <b>←</b> : | | ==X= | ==== | => | X | |

# 10.2.1.2. Part B (Cohorts 2-5)

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | Study Period (Days) | | | | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| Outpatient Visit | Х | | | | | | | | | | | | | | | | | | | Х | |
| Admission to Clinical Unit | | Х | | | | | | | | | | | | | | | | | | | |
| Inpatient Stay at<br>Clinical Unit | | | <b>←=</b> : | ==== | ==== | | ====: | | ==== | ==== | X=== | ==== | ===== | ==== | ==== | | ==== | ==> | | | |
| Discharge from<br>Clinical Unit | | | | | | | | | | | | | | | | | | | х | | Following completion of all assessments. |
| Informed Consent | Х | | | | | | | | | | | | | | | | | | | | |
| Inclusion and Exclusion Criteria | Х | | | | | | | | | | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | | | | | | | | | | | |
| Full Physical<br>Examination | Х | | | | | | | | | | | | | | | | | | Х | | Additional exams/screens |
| Brief Physical<br>Examination | | х | | Х | | х | | | Х | | | Х | | | | | Х | | | Х | may be<br>performed, or<br>brief exams<br>made full<br>exams, by the |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | |
| | | | | | | | | | | | | | | | | | | | | Investigator, as deemed necessary (e.g. where safety or laboratory findings indicate). Tests will be conducted within site specified standards. |
| Height | X | | | | | | | | X | | | | | | | | | | X | |
| Weight Drug/Alcohol/Smoking Screen | X | Х | | | | | | | ٨ | | | | | | | | | | X | Tests include<br>alcohol breath<br>test, smoking<br>breath test and<br>urine drug<br>screen. |
| Medical/Medication/<br>Drug/Alcohol History<br>HIV, Hepatitis B and<br>C Screening | X<br>X | | | | | | | | | | | | | | | | | | | JOI GG11. |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| Tuberculosis Test | Х | | | | | | | | | | | | | | | | | | | | |
| Anti-Nuclear Antibody | X | | | | | | | | Х | | | | | | | | | | Х | | |
| Serum Pregnancy<br>Test (WOCBP only) | Х | | | | | | | | | | | | | | | | | | | Х | |
| Urine Pregnancy Test (WOCBP only) | | Χ | | | | | | | | | | | | | | | | | Х | | |
| Highly effective contraceptive method (WOCBP only) | X | X | Х | Х | X | X | X | X | X | X | Х | X | Х | X | X | X | X | X | X | Х | Must use method for a minimum of 28 days prior to first dose of study medication until the follow- up visit. |
| Contraception with male condoms (WOCBP using hormonal contraceptive method and male subjects with female partners of childbearing potential only) | | Х | X | X | Х | х | Х | X | Х | X | X | X | X | Х | х | Х | Х | X | х | Х | |
| C-SSRS | Χ | <b>←</b> | X→ | | | | | | Χ | | | | | | | | | | Χ | Χc | May be |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | completed on either Day -1 or Day 1, but no later than 1hr prior to dosing. To be completed predose on Day 7. C-SSRS to be conducted on follow-up only in the instance that a subject withdraws from the study. |
| Meals | | x | Х | х | Х | Χ | Χ | X | X | Х | Х | X | X | Х | X | X | Х | Х | X | | TID Dosing: On Day 1 through 14 subjects will fast 8hr overnight. Breakfast will be served approximately |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | 2hr after dosing on Days 1-8, 10, 12 and 13 and 2hr after dosing on Day 14. A "standard" and a "high fat" breakfast will be served approximately 30 minutes prior to dosing on Day 9 and Day 11, respectively. On all study days, lunch and dinner will be served between 2 to 3hr prior to dose 2 and dose 3, |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | respectively. BID Dosing: On Day 1 through 14, subjects will fast 8hr overnight prior to dose 1. A breakfast will be served approximately 2hr after dose 1. Lunch will be served approximately 4-5hr after dose 1. Dinner will be served between 2-3hr prior to dose 2. A snack may be consumed approximately 2-3hr after dose 2. |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | Water is permitted with dosing and at all times. Subjects will receive standardized meals scheduled at the same time in each period. Meals will be served as per the site schedule on Days -1, 16 and 17. |
| Haem/Chem/<br>Urinalysis Test<br>(Include Liver<br>Chemistries) | X | Х | х | х | | Х | | | Х | | | Х | | | | | х | | | Х | Collection on<br>Day 1 no later<br>than 1hr prior<br>to dosing. To<br>be drawn pre-<br>dose on Days<br>2, 4, 7 and 10. |
| Fasting lipid panel | Χ | | Χ | Χ | | Χ | | | Χ | | | Χ | | | | | Χ | | | Х | Collection on |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| Holter Monitoring (24-hour) | X | | | | | | | | | | | | | | | | | | | | Day 1 no later<br>than 1hr prior<br>to dosing. To<br>be drawn pre-<br>dose on Days<br>2, 4, 7 and 10. |
| Telemetry | | | ) | ( | ) | ( | | | | | | | | | | ) | < | | | | Continuous at least 24 hr post-evening dose. Initiate at least 15 min. prior to dosing. |
| PK blood sampling | | | Χq | Xe | Xe | Хe | Xe | | Xe | | Χf | | Xf | | | Χg | | | | | d On Day 1, PK<br>samples will<br>be collected<br>pre-dose and<br>at the following<br>time points<br>post first-dose:<br>20min, 40min,<br>1hr, 1hr 30min,<br>2hr, 3hr, 5hr, |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | 7hr, 9hr and 11hr. e On Days 2,3 4, 5 and 7 predose samples only. f Days 9, and 11: Cohort 2, 3 and Cohort 4 PK sampling will be collected predose and at the following time points post first-dose: 20min, 40min, 1hr, 1hr 30min, 2hr, 3hr, 5hr, 7hr (prior to 2nd dose) 7hr 20min, 7hr 40 min, 8hr, 8hr 30min, 9hr, 10hr, 12hr. |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | Cohort 5 is currently not planned to have PK assessment but may be included depending on outcome of food effect in Cohorts 2, 3 and 4. 9 Day 14 sampling for Cohorts 2, 3, 4 and 5 will be over 24hr according to the following schedules: For <u>TID</u> <u>Dosing:</u> PK samples to be taken pre-dose and then at the |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | following time points post first-dose: 20min, 40min, 1hr, 1hr 30min, 2hr, 3hr, 5hr, 7hr (pre-2nd dose) 7hr 20min, 7hr 40 min, 8hr, 8hr 30min, 9hr, 10hr, 12hr, 14hr (pre 3rd dose), 14hr 20min, 15hr, 15hr 30min, 16hr, 17hr, 19hr, 22hr, 24hr. For BID Dosing: PK samples to be taken pre-dose on Day 1 and then at the |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | subsequent time points post first-dose: 20min, 40min, 1hr, 1hr 30min, 2hr, 3hr, 4hr, 6hr, 8hr, 10hr, 12hr (pre 2nd dose), 12hr 20min, 12hr 40min, 13hr, 13hr 30min, 14hr, 15hr, 16hr, 19hr, 22hr, 24hr. |
| Metabolite sampling | | | | | | | | | | | | | | | | Xh | | | | | h Metabolite<br>sampling will<br>be conducted<br>pre-dose and<br>2hr post first<br>dose on Day<br>14 only. |
| 4β-hydroxycholesterol sampling | | | Xi | | | | | | | | | | | | | | Хi | | | | <sup>i</sup> Sample to be<br>taken pre-dose<br>on Day 1 in a |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | fasted state. Sample to be taken at 24hr post first dose on Day 14. Sample should be in a fasted state. TID Dosing: |
| Neuro. examination | | | X | X | X | | | | X | | | | | | | | | X | | | Neurological examinations to be conducted either on Day-1 or pre-dose Day 1 and then at the subsequent time points post first dose: 2hr, 9hr, 16hr, 24hr and 48hr. To be completed pre-dose on Day 7 |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | and then 48 hr post-last dose on Day 14. BID Dosing: Neurological examinations to be conducted predose either on Day-1 or Day 1 and then at the subsequent time points post first dose: 2hr, 14hr, 24hr and 48hr. To be completed pre-dose on Day 7 and then 48hr post-last dose on Day 14. |
| 12-Lead ECG | Х | Χ | Τ | Χ | | Χ | | | Χ | | | | | | | Χ | | | | Х | Vital signs to |
| Vital signs | X | Χ | Т | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | include HR,<br>BP, |
| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | Study Period (Days) | | | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|--|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | temperature and respiration rate. On Day 1: TID Dosing: 12-Lead ECG and Vital Signs to be conducted on Day-1 and predose Day 1 and then at the subsequent time points post first-dose: 40min, 2hr, 4hr, 7hr (pre-2nd dose), 9hr, 14hr (pre-3rd dose), 16hr, 24hr, 48hr. Then 24 and 48hr after the first dose and last dose |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | administered on Day 14. BID Dosing: 12-Lead ECG and Vital Signs to be conducted predose either on Day-1 or Day 1 and then at the subsequent time points post first-dose: 40 min, 2hr, 4hr, 12hr (predose), 14hr, 24hr, 48hr. Then 24 and 48hr after the first and last dose administered on Day 14. On Days 3 to 14, pre-dose |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | samples only.<br>T = Triplicate. |
| Randomization | | | X | | | | | | | | | | | | | | | | | | Randomization<br>can occur on<br>either Day -1<br>or Day 1. |
| Study Treatment | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | TID dosing: GSK2982772 or placebo will be administered using a 7hr, 7hr and 10hr dosing interval. BID dosing: GSK2982772 or placebo will be administered using a 12hr dosing interval. |
| Pharmacogenetic<br>Sample (PGx) | | | Х | | | | | | | | | | | | | | | | | | A PGx blood<br>sample is<br>collected at the<br>Day 1 visit, |

| Procedure | Screening<br>(Up to 28<br>days<br>before<br>Day 1) | | | | | | | | Stu | dy Pe | riod ( | Days) | | | | | | | | Follow-<br>up<br>(No<br>more<br>than 14<br>days<br>post<br>last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -<br>1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | | |
| | | | | | | | | | | | | | | | | | | | | | after the subject has been randomized and provided informed consent for genetic research. If the sample is not collected on Day 1, it can be collected at any time during the study after randomization. |
| AE review | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | |
| SAE review | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | |
| Concomitant medication review | Х | Χ | Χ | Χ | Х | Х | Х | Х | Χ | Χ | Х | Χ | Χ | Х | Χ | Χ | Х | Χ | Х | X | |

### 10.3. Appendix 3: Assessment Windows

### 10.3.1. Definitions of Assessment Windows for Analyses

No Assessment Windows will be defined for Analysis, and summaries and analyses will be based on nominal visits.

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

#### 10.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the start and/or stop date/time of the study treatment within the period for Part A and the start and/or stop date/time of the study treatment for Part B.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date/Time ≤ Study Treatment Start Date/Time |
| On-Treatment | Study Treatment Start Date/Time < Date/Time ≤ Study Treatment Stop Date/Time |
| Post-Treatment | Date/Time > Study Treatment Stop Date/Time |

#### 10.4.1.1. Study Phases for Concomitant Medications

| Treatment State | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing

#### 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date +1. |
| | <ul> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 1 days.</li> </ul> |
| | <ul> <li>For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period it would be counted in both periods. For the initial period the logic would be as above. For the later period the logic would use the treatment dates associated with the later period:</li> </ul> |
| | Treatment Period Start Date ≤ AE Worsening Date ≤ Study Treatment Stop Date + 1 days. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be Treatment Emergent.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

### 10.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Compound | One reporting effort will be set up for this study which combines Part A and Part B: \arenv\arprod\gsk2982772\mid205184\final_01 |
| Analysis Datasets | |
| Analysis datasets will be created according to Integrated Data Standards Library (IDSL) GSK A&R dataset standards | |
| Generation of RTF Files | |
| RTF files will be generated for all tables within the final_01 reporting effort. | |

#### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All participant level listings should be located in the modular appendices as ICH or non-ICH listings.
- All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### **Formats**

- All data will be reported according to the actual treatment the participant received, unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables and figures:
  - Planned time relative to dosing will be used in figures and summaries and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).

| Unscheduled | <ul> <li>Unscheduled or unplanned readings will be presented within the participant's listings.</li> </ul> |
|---|---|
| Unscheduled Visits | |
| <ul> <li>Unscheduled visits</li> </ul> | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled vis | All unscheduled visits will be included in listings. |
| <b>Descriptive Summary</b> | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to PKOne. Note: Concentration values will be imputed as per GUI_51487. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Parameter Derivation | |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: $C_0$ , $C_7$ , $C_{12}$ , $C_{14}$ , $C_{24}$ . |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to PKOne. |

#### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented except for blood pressure measurements as only the average of the 3 blood pressure readings will be recorded on the CRF.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → S
- $\rightarrow$  Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### 10.6.2. Study Population

#### **Date of Birth**

Only the year of birth will be captured, and therefore the date of birth is then derived as follows:
 Year of birth = YYYY → Date of birth = 30th June YYYY

#### Age

- •
- Calculated as the integer part of (date of screening date of birth)

Age = integer part (date of screening – 30<sup>th</sup> June YYYY) / 365.25.

Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m) 2]

#### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

- Frequency is 2 for BID and 3 for TID. Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is defined as 1 day in Part A in each period and 14 days in Part B.

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### 10.6.3. Safety

#### **ECG Parameters**

#### **RR Interval**

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - If QTcF is machine read, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcF will be derived as:

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

# 10.7. Appendix 7: Reporting Standards for Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the last scheduled procedure shown in the SoA (see Appendix 2).</li> <li>Withdrawn participants may be replaced in the study. Additional replacement participants may be randomized to guarantee that sufficient participants are treated with GSK2982772 at any given dose before escalating to the following dose. Replacement participants will be assigned to the same treatment sequence (Cohort 1) or treatment (Cohorts 2-5) but have different subject numbers and randomisation numbers assigned.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |
| Liver<br>Chemistry<br>Stopping<br>Criteria | <ul> <li>Discontinuation of study treatment for abnormal liver tests is required when: <ul> <li>in the presence of abnormal liver chemistries not meeting protocol-specified stopping rules, the investigator believes study treatment discontinuation is in the best interest of the participant.</li> <li>ALT ≥ 3 x ULN.</li> </ul> </li> <li>Note: Refer to Appendix 7 of the protocol for details of the required assessments if a participant meets the above criteria.</li> </ul> |
| QTc<br>Stopping<br>Criteria | A participant that meets either bulleted criterion based on the average of triplicate ECG readings will be withdrawn from study treatment: |
| Nervous<br>System<br>Stopping<br>Criteria | <ul> <li>A participant will be withdrawn from the study if: <ul> <li>A Grade 3 or greater CTCAE Nervous System finding is observed or a significant neurologic change from a participant's baseline physical examination is observed.</li> <li>Any adverse event included in the CTCAE for Nervous System, which is also considered to be clinically significant by the Principal Investigator, will be reviewed for potential participant withdrawal.</li> </ul> </li> </ul> |

### 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from </li> </ul> |
| | the table. o Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such. |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.8. Appendix 8: Values of Potential Clinical Importance

# 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | D. ". ( | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | ' | $\Delta$ from BL | ↓0.075 | |
| | g/L | Male | | 180 |
| Haemoglobin | | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

### 10.8.2. ECG

| ECG Parameter | Units | Category | Clinical Concern Range | |
|---|---|---|---|---|
| | | | Lower | Upper |
| Absolute | | | | |
| | msec | H1 | > 450 | < 480 |
| Absolute QTc Interval | | H2 | ≥ 480 | < 500 |
| | | Н3 | ≥ 500 | |
| Absolute PR Interval | msec | L, H | < 110 | > 220 |
| Absolute QRS Interval | msec | L, H | < 75 | > 110 |
| Change from Baseline | | | | |
| Increase from Baseline | mcoo | H1 | > 30 | ≤ 59 |
| QTc | msec | H2 | ≥ 60 | |

# 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |
| Respiratory Rate | breaths/min | ≤ 8 | ≥ 20 |
| Temperature | °C | ≤ 35.5 | ≥37.8 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

# 10.9. Appendix 9: Abbreviations & Trade Marks

### 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ALT | Alanine aminotransferase |
| A&R | Analysis and Reporting |
| AUC | AUC Area under the concentration-time curve |
| AUC(0-7) | Area under the concentration-time curve from time zero to 7 hours post first |
| , | dose (TID dosing) |
| AUC(7-14) | Area under the concentration-time curve from 7 to 14 hours post first dose |
| , , | (TID dosing) |
| AUC(14-24) | Area under the concentration-time curve from 14 to 24 hours post first dose |
| | (TID dosing) |
| AUC(0-12) | Area under the concentration-time curve from 0 to 12 hours post first dose |
| | (BID dosing) |
| AUC(12-24) | Area under the concentration-time curve from 12 to 24 hours post first dose |
| | (BID dosing) |
| AUC(0-24) | Area under the concentration-time curve from time zero to 24 hours post |
| | first dose |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to last |
| | time of quantifiable concentration within a participant across all treatments |
| AUC(0-т) | AUC from 0 hours to the time of next dosing |
| BID | Twice a day |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |

| Abbreviation | Description |
|---|---|
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Friderica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SoA | Schedule of Activities |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TID | Three times a day |
| Tmax | Time taken to maximum observed plasma drug concentration |

#### 10.9.2. Trademarks

| | ks of the GlaxoSmithKline oup of Companies |
|------|--------------------------------------------|
| HARP | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

#### 10.10. Appendix 10: List of Data Displays

#### 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-----------------------|------------|
| Study Population | 1.1 to 1.23 | N/A |
| Safety | 2.1 to 2.41 | 2.1 to 2.6 |
| Pharmacokinetic | 3.1 to 3.10 | 3.1 to 3.8 |
| Section | List | ings |
| ICH Listings | 1 to 33 and 40 to 73 | |
| Other Listings | 34 to 39 and 74 to 79 | |

#### 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------|---------|---------|
| Study Population | N/A | N/A | N/A |
| Safety | N/A | SAFE_T1 | SAFE_L1 |
| Pharmacokinetic | N/A | N/A | N/A |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 10.10.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | Cohort 1 - sing | gle ascending dos | e, 3-way crossover): Subject Disposition | | |
| 1.1. | Safety<br>(Part A) | ES1A | Summary of Subject Disposition for the Subject Conclusion Record (Part A) | ICH E3, FDAAA, EudraCT Add footnote: Note: "Subjects" is used to refer to "Participants" in all data displays to reflect GSK display standards and CDISC SDTM/ADaM standards. | SAC |
| 1.2. | Safety<br>(Part A) | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment (Part A) | ICH E3 | SAC |
| 1.3. | Safety<br>(Part A) | ES4 | Summary of Disposition at Each Study Epoch (Part A) | ICH E3 | SAC |
| 1.4. | All Subject<br>(Part A) | ES6 | Summary of Screening Status and Reasons for Screen Failure (Part A) | Journal Requirements | SAC |
| Part A | Part A (Cohort 1 – single ascending dose, 3-way crossover): Protocol Deviation | | | | |
| 1.5. | Safety<br>(Part A) | DV1 | Summary of Important Protocol Deviations (Part A) | ICH E3 | SAC |

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | (Cohort 1 – sin | gle ascending dos | se, 3-way crossover): Population Analysed | • | |
| 1.6. | All Subjects<br>(Part A) | SP1 | Summary of Study Populations (Part A) | IDSL Add the following footnotes: [1] Subjects are included in the Randomised population if they were randomly assigned to treatment in the study. [2] Subjects are included in the Safety population if they have been randomized and received at least one dose of study treatment. [3] Subjects are included in the Pharmacokinetic population if they are in the Safety Population and a pharmacokinetic sample was obtained and analysed. | SAC |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): Demographic and Baseline Characteristi | cs | |
| 1.7. | Safety<br>(Part A) | DM3 | Summary of Demographic Characteristics (Part A) | ICH E3, FDAAA, EudraCT Do not include Weight (to be included in Vital Signs summary) Add Footnote: [1] For calculating age, birth date is imputed as June 30 in the year of birth. | SAC |

| Study F | Population Tabl | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.8. | Randomised<br>(Part A) | DM11 | Summary of Age Ranges (Part A) | EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years')) Please add footnote to say that randomised population=enrolled population. | SAC |
| 1.9. | Safety<br>(Part A) | DM5 | Summary of Race and Racial Combinations (Part A) | ICH E3, FDA, FDAAA, EudraCT | SAC |
| Part A | Cohort 1 – sing | gle ascending dos | e, 3-way crossover): Medical Conditions and Prior and Concor | nitant Medications | |
| 1.10. | Safety<br>(Part A) | MH1 /<br>MH4 | Summary of Current/Past Medical Conditions (Part A) | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.11. | Safety<br>(Part A) | CM1 | Summary of Concomitant Medications (Part A) | ICH E3 | SAC |
| Part A | Cohort 1 – sing | gle ascending dos | e, 3-way crossover): Exposure and Treatment Compliance | | |
| 1.12. | Safety<br>(Part A) | EX5 | Summary of Exposure to Study Treatment (Part A) | ICH E3 Total daily dose (mg) and number of days | SAC |
| Part B | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Subject Disposition | · | |
| 1.13. | Safety<br>(Part B) | ES1 | Summary of Subject Disposition for the Subject Conclusion Record (Part B) | ICH E3, FDAAA, EudraCT | SAC |
| 1.14. | Safety<br>(Part B) | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment (Part B) | ICH E3 | SAC |

| Study F | opulation Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.15. | All Subjects<br>(Part B) | ES6 | Summary of Screening Status and Reasons for Screen Failure (Part B) | Journal Requirements | SAC |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | ose, sequential-group): Protocol Deviation | | |
| 1.16. | Safety<br>(Part B) | DV1 | Summary of Important Protocol Deviations (Part B) | ICH E3 | SAC |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | ose, sequential-group): Population Analysed | | |
| 1.17. | Safety<br>(Part B) | SP1 | Summary of Study Populations (Part B) | IDSL Add the following footnotes: [1] Subjects are included in the Randomised population if they were randomly assigned to treatment in the study. [2] Subjects are included in the Safety population if they have been randomized and received at least one dose of study treatment. [3] Subjects are included in the Pharmacokinetic population if they are in the Safety Population and a pharmacokinetic sample was obtained and analysed. | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Demographic and Baseline Characterist | tics | |
| 1.18. | Safety<br>(Part B) | DM1 | Summary of Demographic Characteristics (Part B) | ICH E3, FDAAA, EudraCT Do not include Weight (to be included in Vital Signs summary) [1] For calculating age, birth date is imputed as June 30 in the year of birth. | SAC |
| 1.19. | Randomised<br>(Part B) | DM11 | Summary of Age Ranges (Part B) | EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years')) | SAC |
| 1.20. | Safety<br>(Part B) | DM5 | Summary of Race and Racial Combinations (Part B) | ICH E3, FDA, FDAAA, EudraCT | SAC |
| Part B | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Medical Conditions and Prior and Conc | omitant Medications | |
| 1.21. | Safety<br>(Part B) | MH1 /<br>MH4 | Summary of Current/Past Medical Conditions (Part B) | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.22. | Safety<br>(Part B) | CM1 | Summary of Concomitant Medications (Part B) | ICH E3 | SAC |
| Part B | (Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Exposure and Treatment Compliance | | |
| 1.23. | Safety<br>(Part B) | EX1 | Summary of Exposure to Study Treatment (Part B) | ICH E3 Total daily dose, cumulative actual dose and number of days. | SAC |

# 10.10.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): Adverse Events (AEs) | | |
| 2.1. | Safety<br>(Part A) | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Part A) | | SAC |
| 2.2. | Safety<br>(Part A) | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Part A) | ICH E3 | SAC |
| 2.3. | Safety<br>(Part A) | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity (Part A) | ICH E3 | SAC |
| 2.4. | Safety<br>(Part A) | AE15 | Summary of Common (>=10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) (Part A) | FDAAA, EudraCT | SAC |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): Serious and Other Significant Adverse Ev | rents | |
| 2.5. | Safety<br>(Part A) | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) (Part A) | FDAAA, EudraCT Only if 3 or more SAEs reported | SAC |
| 2.6. | Safety<br>(Part A) | AE3 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Overall Frequency (Part A) | IDSL | SAC |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): Laboratory: Chemistry | | |
| 2.7. | Safety<br>(Part A) | LB1 | Summary of Chemistry Changes from Baseline (Part A) | ICH E3 | SAC |
| 2.8. | Safety<br>(Part A) | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline (Part A) | ICH E3 | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.9. | Safety<br>(Part A) | LB17 | Summary of Worst Case Lipids Outside Laboratory Normal Range Post-Baseline Relative to Baseline (Part A) | | SAC |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): Laboratory: Hematology | <u> </u> | • |
| 2.10. | Safety<br>(Part A) | LB1 | Summary of Hematology Changes from Baseline (Part A) | ICH E3 | SAC |
| 2.11. | Safety<br>(Part A) | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline (Part A) | ICH E3 | SAC |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): Laboratory: Urinalysis | | • |
| 2.12. | Safety<br>(Part A) | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Part A) | ICH E3 | SAC |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): Laboratory: Hepatobiliary (Liver) | | |
| 2.13. | Safety<br>(Part A) | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting (Part A) | IDSL | SAC |
| 2.14. | Safety<br>(Part A) | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities (Part A) | IDSL | SAC |
| Part A | (Cohort 1 – sing | gle ascending dos | se, 3-way crossover): ECG | | |
| 2.15. | Safety<br>(Part A) | EG1 | Summary of ECG Findings (Part A) | IDSL | SAC |
| 2.16. | Safety<br>(Part A) | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category (Part A) | IDSL | SAC |
| 2.17. | Safety<br>(Part A) | EG2 | Summary of Change from Baseline in ECG Values by Visit (Part A) | IDSL | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18. | Safety<br>(Part A) | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category (Part A) | IDSL | SAC |
| Part A | Cohort 1 – sing | gle ascending dos | e, 3-way crossover): Vital Signs | | • |
| 2.19. | Safety<br>(Part A) | VS1 | Summary of Change from Baseline in Vital Signs (Part A) | ICH E3 | SAC |
| Part A | Cohort 1 – sinç | gle ascending dos | e, 3-way crossover): Suicide Risk Monitoring | | • |
| 2.20. | Safety<br>(Part A) | CSSRS1 | Summary of Subjects with C-SSRS Suicidal Ideation or Behaviour during Treatment (Part A) | | SAC |
| Part B | (Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Adverse Events (AEs)) | | |
| 2.21. | Safety<br>(Part B) | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Part B) | ICH E3 | SAC |
| 2.22. | Safety<br>(Part B) | AE3 | Summary of Common (>=10%) Adverse Events by Overall Frequency (Part B) | ICH E3 | SAC |
| 2.23. | Safety<br>(Part B) | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity (Part B) | ICH E3 | SAC |
| 2.24. | Safety<br>(Part B) | AE15 | Summary of Common (>=10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subject and Occurrences) (Part B) | FDAAA, EudraCT | SAC |
| Part B | (Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Serious and Other Significant Adverse l | Events | |
| 2.25. | Safety<br>(Part B) | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) (Part B) | FDAAA, EudraCT Only if 3 or more SAEs reported | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.26. | Safety<br>(Part B) | AE3 | Summary of Adverse Events Leading to Permanent<br>Discontinuation of Study Treatment or Withdrawal from Study by<br>Overall Frequency (Part B) | IDSL | SAC |
| Part B | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Laboratory: Chemistry | | |
| 2.27. | Safety<br>(Part B) | LB1 | Summary of Chemistry Changes from Baseline (Part B) | ICH E3 | SAC |
| 2.28. | Safety<br>(Part B) | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline (Part B) | ICH E3 | SAC |
| 2.29. | Safety<br>(Part A) | LB17 | Summary of Worst Case Lipids Outside Laboratory Normal Range Post-Baseline Relative to Baseline (Part B) | | SAC |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Laboratory: Hematology | | |
| 2.30. | Safety<br>(Part B) | LB1 | Summary of Hematology Changes from Baseline (Part B) | ICH E3 | SAC |
| 2.31. | Safety<br>(Part B) | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline (Part B) | ICH E3 | SAC |
| Part B | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Laboratory: Urinalysis | | |
| 2.32. | Safety<br>(Part B) | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Part B) | ICH E3 | SAC |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Laboratory: Hepatobiliary (Liver) | | |
| 2.33. | Safety<br>(Part B) | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting (Part B) | IDSL | SAC |
| 2.34. | Safety<br>(Part B) | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities (Part B) | IDSL | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Laboratory: Other | | |
| 2.35. | Pharmacoki<br>netic<br>(Part B) | Non-Standard<br>SAFE_T1 | Summary of Plasma 4β-hydroxycholesterol to Cholesterol Ratio (Part B) | Include SE and 95% CI. | SAC |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | ose, sequential-group): ECG | | |
| 2.36. | Safety<br>(Part B) | EG1 | Summary of ECG Findings (Part B) | IDSL | SAC |
| 2.37. | Safety<br>(Part B) | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category (Part B) | IDSL | SAC |
| 2.38. | Safety<br>(Part B) | EG2 | Summary of Change from Baseline in ECG Values by Visit (Part B) | IDSL | SAC |
| 2.39. | Safety<br>(Part B) | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category (Part B) | IDSL | SAC |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Vital Signs | | |
| 2.40. | Safety<br>(Part B) | VS1 | Summary of Change from Baseline in Vital Signs (Part B) | ICH E3 | SAC |
| Part B ( | Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Suicide Risk Monitoring | | |
| 2.41. | Safety<br>(Part B) | CSSRS1 | Summary of Subjects with C-SSRS Suicidal Ideation or Behaviour during Treatment (Part B) | | SAC |

# 10.10.6. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | (Cohort 1 – sin | gle ascending dos | e, 3-way crossover): Adverse Events | | |
| 2.1. | Safety<br>(Part A) | AE10 | Plot of Common (>=10%) Adverse Events and Relative Risk (Part A) | IDSL<br>Common defined as >10% | SAC |
| Part A | (Cohort 1 – sin | gle ascending dos | e, 3-way crossover): Hepatobiliary (Liver) | | |
| 2.2. | Safety<br>(Part A) | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT (Part A) | | SAC |
| 2.3. | Safety<br>(Part A) | LIVER9 | Scatter Plot for Maximum ALT vs. Maximum Total Bilirubin (Part A) | | SAC |
| Part B | (Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Adverse Events | | |
| 2.4. | Safety<br>(Part B) | AE10 | Plot of Common (>=10%) Adverse Events and Relative Risk (Part B) | IDSL<br>Common defined as >10% | SAC |
| Part B | (Cohorts 2, 3, 4 | and 5 - repeat do | se, sequential-group): Hepatobiliary (Liver) | | |
| 2.5. | Safety<br>(Part B) | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT (Part B) | | SAC |
| 2.6. | Safety<br>(Part B) | LIVER9 | Scatter Plot for Maximum ALT vs. Maximum Total Bilirubin (Part B) | | SAC |

#### 10.10.7. Pharmacokinetic Tables

| Pharm | nacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | (Cohort 1 – single a | scending dose, | 3-way crossover): Pharmacokinetic Concentrations | | |
| 3.1. | Pharmacokinetic<br>(Part A) | PK01 | Summary of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data (Part A) | Include column for 95% CI. | SAC |
| 3.2. | Pharmacokinetic<br>(Part A) | PK01 | Summary of Plasma M8 (GSK3562183) Pharmacokinetic Concentration-Time Data (Part A) | Include column for 95% CI. | SAC |
| 3.3. | Pharmacokinetic<br>(Part A) | PK01 | Summary of Plasma M9 (GSK2997852) Pharmacokinetic Concentration-Time Data (Part A) | Include column for 95% CI. | SAC |
| Part A | (Cohort 1 – single a | scending dose, | 3-way crossover): Pharmacokinetic Parameters | | |
| 3.4. | Pharmacokinetic<br>(Part A) | PK03 | Summary of Derived Plasma GSK2982772 Pharmacokinetic Parameters (Part A) | Include columns for parameter, period, treatment, N, n, mean, 90% CI, standard deviation [SD], standard error [SE], median, minimum and maximum. | SAC |
| 3.5. | Pharmacokinetic<br>(Part A) | PK05 | Summary of Log-Transformed Derived Plasma GSK2982772<br>Pharmacokinetic Parameters (Part A) | Include columns for parameter, period, treatment, N, n, geometric mean, 90% CI of geometric mean, standard deviation [SD] of logged data and %CVb. Do not summarise Tmax. | SAC |
| Part B | (Cohorts 2, 3, 4 and | 5 - repeat dose | e, sequential-group): Pharmacokinetic Concentrations | 20 Het dammando Tinaxi | |
| 3.6. | Pharmacokinetic<br>(Part B) | PK01 | Summary of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data (Part B) | Include column for 95% CI and the SE. | SAC |

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.7. | Pharmacokinetic<br>(Part B) | PK01 | Summary of Plasma M8 (GSK3562183) Pharmacokinetic Concentration-Time Data (Part B) | Include column for 95% CI and the SE. | SAC |
| 3.8. | Pharmacokinetic<br>(Part B) | PK01 | Summary of Plasma M9 (GSK2997852) Pharmacokinetic Concentration-Time Data (Part B) | Include column for 95% CI and the SE. | SAC |
| Part B | (Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): Pharmacokinetic Parameters | | |
| 3.9. | Pharmacokinetic<br>(Part B) | PK03 | Summary of Derived Plasma GSK2982772 Pharmacokinetic Parameters (Part B) | Include columns for parameter, treatment, N, day, fed/fasted state, n, mean, 90% CI, standard deviation [SD], SE, median, minimum and maximum. | SAC |
| 3.10. | Pharmacokinetic<br>(Part B) | PK05 | Summary of Log-Transformed Derived Plasma GSK2982772<br>Pharmacokinetic Parameters (Part B) | Include columns for parameter, treatment, N, day, fed/fasted state, n, geometric mean, 90% CI of geometric mean, standard deviation [SD] of logged data and %CVb. Do not summarise Tmax. | SAC |

# 10.10.8. Pharmacokinetic Figures

| Pharm | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | (Cohort 1 – single a | scending dose, | 3-way crossover): Pharmacokinetic Concentrations | | |
| 3.1. | Pharmacokinetic<br>(Part A) | PK16b | Individual Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) (Part A) | | SAC |
| 3.2. | Pharmacokinetic<br>(Part A) | PK24 | Individual Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) by Treatment (Part A) | | SAC |
| 3.3. | Pharmacokinetic<br>(Part A) | PK19 | Mean (+ SE) Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) (Part A) | | SAC |
| 3.4. | Pharmacokinetic<br>(Part A) | PK20 | Median (Range) Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) (Part A) | | SAC |
| Part B | (Cohorts 2, 3, 4 and | l 5 – repeat dose | , sequential-group): Pharmacokinetic Concentrations | | |
| 3.5. | Pharmacokinetic<br>(Part B) | PK16a | Individual Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) (Part B) | | SAC |
| 3.6. | Pharmacokinetic<br>(Part B) | PK24 | Individual Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) by Treatment (Part B) | | SAC |
| 3.7. | Pharmacokinetic<br>(Part B) | PK19 | Mean (+ SE) Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) (Part B) | | SAC |
| 3.8. | Pharmacokinetic<br>(Part B) | PK20 | Median (Range) Plasma GSK2982772 Concentration-Time Plots (Linear and Semi-log) (Part B) | | SAC |

# 10.10.9. ICH Listings

| ICH: Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Subject Disposition | | |
| 1. | All Subjects<br>(Part A) | ES7 | Listing of Reasons for Screen Failure (Part A) | Journal Guidelines | SAC |
| 2. | Safety<br>(Part A) | ES3 | Listing of Reasons for Study Withdrawal (Part A) | ICH E3 | SAC |
| 3. | Safety<br>(Part A) | SD3 | Listing of Reasons for Study Treatment Discontinuation (Part A) | ICH E3 | SAC |
| 4. | Safety<br>(Part A) | BL2 | Listing of Subjects for Whom the Treatment Blind was Broken (Part A) | ICH E3 | SAC |
| 5. | Safety<br>(Part A) | TA1 | Listing of Planned and Actual Treatments (Part A) | IDSL | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Protocol Deviations | | 1 |
| 6. | Safety<br>(Part A) | DV2A | Listing of Important Protocol Deviations (Part A) | ICH E3 | SAC |
| 7. | Safety<br>(Part A) | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Part A) | ICH E3 | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Populations Analysed | | |
| 8. | All Subjects<br>(Part A) | SP3a | Listing of Subjects Excluded from Any Population (Part A) | ICH E3 | SAC |

| ICH: Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Demographic and Baseline Characteristics | | |
| 9. | Safety<br>(Part A) | DM4 | Listing of Demographic Characteristics (Part A) | ICH E3 Do not include Weight. | SAC |
| 10. | Safety<br>(Part A) | DM10 | Listing of Race (Part A) | ICH E3 | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Prior and Concomitant Medications | | • |
| 11. | Safety<br>(Part A) | CP_CM4 | Listing of Concomitant Medications (Part A) | IDSL | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Exposure and Treatment Compliance | | • |
| 12. | Safety<br>(Part A) | EX4 | Listing of Exposure Data (Part A) | ICH E3 | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Adverse Events | | • |
| 13. | Safety<br>(Part A) | AE9CP | Listing of All Adverse Events (Part A) | ICH E3 | SAC |
| 14. | Safety<br>(Part A) | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part A) | ICH E3 | SAC |
| 15. | Safety<br>(Part A) | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text (Part A) | IDSL | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Serious and Other Significant Adverse Ever | nts | |
| 16. | Safety<br>(Part A) | AE9CPa | Listing of Serious Adverse Events (Part A) | ICH E3 Include fatal and non-fatal status | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 17. | Safety<br>(Part A) | AE14 | Listing of Reasons for Considering as a Serious Adverse Event (Part A) | ICH E3 | SAC |
| 18. | Safety<br>(Part A) | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment (Part A) | ICH E3 Include fatal and non-fatal status | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Hepatobiliary (Liver) | | |
| 19. | Safety<br>(Part A) | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events (Part A) | IDSL | SAC |
| 20. | Safety<br>(Part A) | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part A) | IDSL | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): All Laboratory | | |
| 21. | Safety<br>(Part A) | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance (Part A) | ICH E3 | SAC |
| 22. | Safety<br>(Part A) | LB6 | Listing of Laboratory Values of Potential Clinical Importance (Part A) | | SAC |
| 23. | Safety<br>(Part A) | LB6 | Listing of All Lipid Data for Subjects with Any Value outside of Laboratory Normal Range (Part A) | Please include additional column after Lab Param for fasting status (if present) | SAC |
| 24. | Safety<br>(Part A) | LB14 | Listing of Laboratory Data with Character Results (Part A) | ICH E3 | SAC |
| 25. | Safety<br>(Part A) | UR2B | Listing of All Urinalysis Data for Subjects with Any Value of Potential Clinical Importance (Part A) | ICH E3 | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): ECG | | |
| 26. | Safety<br>(Part A) | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance (Part A) | IDSL Include absolute PCI subjects. Footnote: Note: H= High absolute value, L= Low absolute value. For QTc Interval H1= >450msec and <480msec, H2= >=480msec and <500msec, H3= >=500msec. | SAC |
| 27. | Safety<br>(Part A) | EG4 | Listing of All ECG Changes for Subjects with Any Change of Potential Clinical Importance (Part A) | Include change from baseline PCI subjects. Footnote: Note: H=High change from baseline value, L=Low change from baseline value. For QTc Interval H1= >30msec and <=59msec, H2= >=60msec | SAC |
| 28. | Safety<br>(Part A) | EG4 | Listing of ECG Values of Potential Clinical Importance (Part A) | IDSL Include absolute PCIs. Footnote: Note: H=High absolute value, L=Low absolute value. For QTc Interval H1= >450msec and <480msec, H2= >=480msec and <500msec, H3= >=500msec. | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 29. | Safety<br>(Part A) | EG4 | Listing of ECG Changes of Potential Clinical Importance (Part A) | Include change from baseline PCIs. Footnote: Note: H=High change from baseline value, L=Low change from baseline value. For QTc Interval H1= >30msec and <=59msec, H2= >=60msec | SAC |
| 30. | Safety<br>(Part A) | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding (Part A) | IDSL | SAC |
| 31. | Safety<br>(Part A) | EG6 | Listing of Abnormal ECG Findings (Part A) | IDSL | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Vital Signs | | |
| 32. | Safety<br>(Part A) | VS5 | Listing of All Vital Signs Values for Subjects with Any Value of Potential Clinical Importance (Part A) | IDSL Footnote: Note: For absolute results: H=High, L=Low. For change from baseline: H1=Lower Increase, H2=Upper Increase, L1=Lower Decrease, L2=Upper Decrease. | SAC |
| 33. | Safety<br>(Part A) | VS5 | Listing of Vital Signs Values of Potential Clinical Importance (Part A) | IDSL Footnote: Note: For absolute results: H=High, L=Low. For change from baseline: H1=Lower Increase, H2=Upper Increase, L1=Lower Decrease, L2=Upper Decrease. | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): Disposition | | |
| 40 | All Subjects<br>(Part B) | ES7 | Listing of Reasons for Screen Failure (Part B) | Journal Guidelines | SAC |
| 41 | Safety<br>(Part B) | ES2 | Listing of Reasons for Study Withdrawal (Part B) | ICH E3 | SAC |
| 42 | Safety<br>(Part B) | SD2 | Listing of Reasons for Study Treatment Discontinuation (Part B) | ICH E3 | SAC |
| 43 | Safety<br>(Part B) | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken (Part B) | ICH E3 | SAC |
| 44 | Safety<br>(Part B) | TA1 | Listing of Planned and Actual Treatments (Part B) | IDSL | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 - repeat dose | , sequential-group): Protocol Deviations | | |
| 45 | Safety<br>(Part B) | DV2 | Listing of Important Protocol Deviations (Part B) | ICH E3 | SAC |
| 46 | Safety (Part B) | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Part B) | ICH E3 | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): Populations Analysed | | |
| 47 | All Subjects<br>(Part B) | SP3 | Listing of Subjects Excluded from Any Population (Part B) | ICH E3 | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): Demographic and Baseline Characteristic | S | |
| 48 | Safety<br>(Part B) | DM2 | Listing of Demographic Characteristics (Part B) | ICH E3 Do not include Weight. | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 49 | Safety<br>(Part B) | DM9 | Listing of Race (Part B) | ICH E3 | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | sequential-group): Prior and Concomitant Medications | | |
| 50 | Safety<br>(Part B) | CP_CM3 | Listing of Concomitant Medications (Part B) | IDSL | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | sequential-group): Exposure and Treatment Compliance | | |
| 51 | Safety<br>(Part B) | EX3 | Listing of Exposure Data (Part B) | ICH E3 | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): Adverse Events | | |
| 52 | Safety<br>(Part B) | AE8CP | Listing of All Adverse Events (Part B) | ICH E3 | SAC |
| 53 | Safety<br>(Part B) | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part B) | ICH E3 | SAC |
| 54 | Safety<br>(Part B) | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text (Part B) | IDSL | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): Serious and Other Significant Adverse Evo | ents | |
| 55 | Safety<br>(Part B) | AE8CPa | Listing of Serious Adverse Events (Part B) | ICH E3 Include fatal and non-fatal status. | SAC |
| 56 | Safety<br>(Part B) | AE14 | Listing of Reasons for Considering as a Serious Adverse Event (Part B) | ICH E3 | SAC |
| 57 | Safety<br>(Part B) | AE8CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment (Part B) | ICH E3 Include fatal and non-fatal status. | SAC |

| ICH: Lis | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B ( | Cohorts 2, 3, 4 and | 5 - repeat dose, | sequential-group): Hepatobiliary (Liver) | | |
| 58 | Safety<br>(Part B) | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events (Part B) | IDSL | SAC |
| 59 | Safety<br>(Part B) | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part B) | IDSL | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 - repeat dose, | sequential-group): All Laboratory | | |
| 60 | Safety<br>(Part B) | LB5 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance (Part B) | ICH E3 | SAC |
| 61 | Safety<br>(Part B) | LB5 | Listing of Laboratory Values of Potential Clinical Importance (Part B) | | SAC |
| 62 | Safety<br>(Part A) | LB6 | Listing of All Lipid Data for Subjects with Any Value outside of Laboratory Normal Range | Please include additional column after Lab Param for fasting status (if present) | SAC |
| 63 | Safety<br>(Part B) | LB14 | Listing of Laboratory Data with Character Results (Part B) | ICH E3 | SAC |
| 64 | Safety<br>(Part B) | UR2A | Listing of All Urinalysis Data for Subjects with Any Value of Potential Clinical Importance (Part B) | ICH E3 | SAC |
| 65 | Pharmacokinetic<br>(Part B) | Non-Standard<br>SAFE_L1 | Listing of Plasma Cholesterol and 4β-hydroxycholesterol Concentration-Time (ug/mL) Data (Part B) | | SAC |

| ICH: Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): ECG | | |
| 66 | Safety<br>(Part B) | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance (Part B) | IDSL Include absolute PCI subjects. Footnote: Note: H= High absolute value, L= Low absolute value. For QTc Interval H1= >450msec and <480msec, H2= >=480msec and <500msec, H3= >=500msec. | SAC |
| 67 | Safety<br>(Part B) | EG3 | Listing of All ECG Changes for Subjects with Any Change of Potential Clinical Importance (Part B) | Include change from baseline PCI subjects. Footnote: Note: H=High change from baseline value, L=Low change from baseline value. For QTc Interval H1= >30msec and <=59msec, H2= >=60msec | SAC |
| 68 | Safety<br>(Part B) | EG3 | Listing of ECG Values of Potential Clinical Importance (Part B) | IDSL Include absolute PCIs. Footnote: Note: H=High absolute value, L=Low absolute value. For QTc Interval H1= >450msec and <480msec, H2= >=480msec and <500msec, H3= >=500msec. | SAC |

| ICH: Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 69 | Safety<br>(Part B) | EG3 | Listing of ECG Changes of Potential Clinical Importance (Part B) | Include change from baseline PCIs. Footnote: Note: H=High change from baseline value, L=Low change from baseline value. For QTc Interval H1= >30msec and <=59msec, H2= >=60msec | SAC |
| 70 | Safety<br>(Part B) | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding (Part B) | IDSL | SAC |
| 71 | Safety<br>(Part B) | EG5 | Listing of Abnormal ECG Findings (Part B) | IDSL | SAC |
| Part B ( | Cohorts 2, 3, 4 and | 5 – repeat dose | , sequential-group): Vital Signs | | |
| 72 | Safety<br>(Part B) | VS4 | Listing of All Vital Signs Values for Subjects with Any Value of Potential Clinical Importance (Part B) | IDSL Footnote: Note: For absolute results: H=High, L=Low. For change from baseline: H1=Lower Increase, H2=Upper Increase, L1=Lower Decrease, L2=Upper Decrease. | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 73 | Safety<br>(Part B) | VS4 | Listing of Vital Signs Values of Potential Clinical Importance (Part B) | IDSL Footnote: Note: For absolute results: H=High, L=Low. For change from baseline: H1=Lower Increase, H2=Upper Increase, L1=Lower Decrease, L2=Upper Decrease. | SAC |

# 10.10.10. Non-ICH Listings

| Non-ICH | l: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Columbia Suicide Severity Rating Scale (C- | SSRS) | |
| 34 | Safety<br>(Part A) | ECSSRS4 | Listing of C-SSRS suicidal Ideation and Behaviour Data (Part A) | | SAC |
| 35 | Safety<br>(Part A) | ECSSRS5 | Listing of C-SSRS Suicidal Behaviour Details (Part A) | | SAC |
| Part A ( | Cohort 1 – single a | scending dose, | 3-way crossover): Pharmacokinetic Data | | |
| 36 | Pharmacokinetic<br>(Part A) | PK08 | Listing of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data (Part A) | | SAC |
| 37 | Pharmacokinetic<br>(Part A) | PK07 | Listing of Plasma M8 (GSK3562183) Pharmacokinetic Concentration-Time Data (Part A) | | SAC |

| Non-ICH | l: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 38 | Pharmacokinetic<br>(Part A) | PK07 | Listing of Plasma M9 (GSK2997852) Pharmacokinetic Concentration-Time Data (Part A) | | SAC |
| 39 | Pharmacokinetic<br>(Part A) | PK14 | Listing of Derived Plasma GSK2982772 Pharmacokinetic Parameters (Part A) | | SAC |
| Part B ( | Cohorts 2, 3, 4 and | l 5 – repeat dose | , sequential-group): Columbia Suicide Severity Rating Scale ( | C-SSRS) | |
| 74 | Safety<br>(Part B) | ECSSRS4 | Listing of C-SSRS suicidal Ideation and Behaviour Data (Part B) | | SAC |
| 75 | Safety<br>(Part B) | ECSSRS5 | Listing of C-SSRS Suicidal Behaviour Details (Part B) | | SAC |
| Part B ( | Cohorts 2, 3, 4 and | l 5 – repeat dose | , sequential-group): Pharmacokinetic Data | | |
| 76 | Pharmacokinetic (Part B) | PK07 | Listing of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data (Part B) | | SAC |
| 77 | Pharmacokinetic (Part B) | PK07 | Listing of Plasma M8 (GSK3562183) Pharmacokinetic Concentration-Time Data (Part B) | | SAC |
| 78 | Pharmacokinetic (Part B) | PK07 | Listing of Plasma M9 (GSK2997852) Pharmacokinetic Concentration-Time Data (Part B) | | SAC |
| 79 | Pharmacokinetic (Part B) | PK13 | Listing of Derived Plasma GSK2982772 Pharmacokinetic Parameters (Part B) | | SAC |

# 10.11. Appendix 11: Example Mock Shells for Data Displays

Example: SAFE\_T1 Page 1 of n

Protocol: 205184

Population: Pharmacokinetic

Table x.x Summary of Plasma 4β-hydroxycholesterol to Cholesterol Ratio (Part B)

Parameter: xxxx

| Treatment | N | Study Day | Planned<br>Relative<br>Time | n | Mean | 95% CI<br>(Lower, Upper) | SD | SE | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 120mg TID | 24 | Day -1/1<br>Day 14 | Pre-dose<br>24 hr | 24<br>23 | XXXX.X<br>XXXX.X | (xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx) | xx.xx<br>xx.xx | xxxx.x<br>xxxx.x | xxxx.x<br>xxxx.x | xxxx<br>xxxx | xxxx<br>xxxx |
| 240mg TID | 24 | Day -1/1<br>Day 14 | Pre-dose<br>24 hr | 24<br>21 | XXXX.X<br>XXXX.X | (xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx) | xx.xx<br>xx.xx | XXXX.X<br>XXXX.X | xxxx.x<br>xxxx.x | XXXX<br>XXXX | XXXX<br>XXXX |
| 360mg BID | 24 | Day -1/1<br>Day 14 | Pre-dose<br>24 hr | 24<br>24 | XXXX.X<br>XXXX.X | (xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx) | XX.XX<br>XX.XX | XXXX.X<br>XXXX.X | XXXX.X<br>XXXX.X | XXXX<br>XXXX | XXXX<br>XXXX |

#### **CONFIDENTIAL**

205184

Page 1 of n Example: SAFE\_L1

Protocol: 205184 Population: Pharmacokinetic

### Table x.x

Listing of Plasma Cholesterol and 4B-hydroxycholesterol Concentration-Time (ug/mL) Data (Part B)

Treatment: XXXXX

| Inv./<br>Subj. | Visit/<br>Date/<br>Study Day | Planned<br>Relative<br>Time | Actual Time | Time<br>Deviation<br>(Hours) | Actual<br>Relative<br>Time | Analyte | Concentration (ug/mL) | Ratio [1] | Excluded from Analysis? [2] |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXXXX | Part B Day 1<br>DDMMMYYYY/<br>1 | Pre-dose | h:mm | -X.XX | -Xh XXm | 4BOH CHOLESTEROL | XXXX.X | XXX.XX | |
| | • | | | | | CHOLESTEROL | XXXX.X | | |
| | Part B Day 14<br>DDMMMYYYY/<br>1 | Pre-dose | h:mm | -X.XX | -Xh XXm | 4BOH CHOLESTEROL | XXXX.X | | |
| | , | | | | | CHOLESTEROL | XXXX.X | | |

<sup>[1]</sup> Plasma 4B-hydroxycholesterol to Cholesterol ratio.[2] Samples excluded from analyses due to >1% haemolysis.